CLINICAL TRIAL: NCT06892054
Title: Sotorasib Combined With First-line Chemotherapy for Advanced Pancreatic Adenocarcinoma With KRAS p.G12C Mutation
Brief Title: Sotorasib Combined With First-line Chemotherapy for Advanced Pancreatic Adenocarcinoma
Acronym: PANSOTO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Apices Soluciones S.L. (Industry); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-24-01; 2024-516233-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-05; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic; sotorasib; TTD-24-01; KRASG12C
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- First-line chemotherapy (gem/nab-P or FOLFIRINOX) combined with sotorasib (Experimental): A minimum of 6 and a maximum of 15 patients will be enrolled to receive first-line chemotherapy (gem/nab-P or mFOLFIRINOX) in combination with sotorasib 960 mg daily (QD).
  The treatment with gem/nab-P and mFOLFIRINOX should be managed as per clinical practice.
  Gem/nab-P and mFOLFIRINOX, are both considered the standard first-line treatment for patients with metastatic disease who have a good performance status.
  Interventions: Drug: Sotorasib, 960 mg, oral daily dose for 4 weeks (28 days)

INTERVENTIONS:
Drug: Sotorasib, 960 mg, oral daily dose for 4 weeks (28 days) — A minimum of 6 and a maximum of 15 patients will be enrolled to receive first-line chemotherapy (gem/nab-P or mFOLFIRINOX) in combination with sotorasib 960 mg daily (QD). The treatment with gem/nab-P and mFOLFIRINOX should be managed as per clinical practice.
  Other Names: Lumykras

SUMMARY:
The main objective of this trial is to evaluate the safety and tolerability of sotorasib combined with first-line chemotherapy for advanced pancreatic adenocarcinoma harboring KRAS p.G12C mutation.

DETAILED DESCRIPTION:
This is a phase 2, multicenter and open-label study of first-line chemotherapy (gemcitabine combined with nab-paclitaxel [gem/nab-P] or modified FOLFIRINOX [mFOLFIRINOX]) in combination with sotorasib for patients with advance pancreatic cancer harboring KRAS p.G12C mutation.The study will be conducted at approximately 25 sites distributed in two countries (Spain and France). The study will consist of a screening period, a treatment period, a safety follow-up (SFU) and long-term follow-up (LTFU) period. A minimum of 6 and a maximum of 15 patients will be enrolled to receive first-line chemotherapy (gem/nab-P or mFOLFIRINOX) in combination with sotorasib 960 mg daily (QD). An interim safety analysis will be conducted by an independent data monitoring committee (DMC) DMC after the first 3 evaluable patients treated with sotorasib combined with gem/nab-P and an additional interim safety analysis with the first 3 evaluable patients treated with sotorasib combined with mFOLFIRINOX have been treated for at least 1 month, respectively. Patients may discontinue treatment because of disease progression, intolerance of treatment leading to treatment discontinuation, initiation of another anticancer therapy, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Men or women aged ≥ 18 years old.
3. Using adequate contraceptive measures or sexual abstinence during the treatment and for 7 additional days after the last dose of sotorasib and for at least 6 months afterwards after the last dose of mFOLFIRINOX or gem/nab-P

   * Female who has been post-menopausal for more than one year or female of childbearing potential using a highly effective method of contraception (i.e., a method with less than 1% failure rate [e.g., sterilization, hormone implants, hormone injections, some intrauterine devices, or vasectomized partner])
   * Male agreeing to use condoms (during the treatment and for 7 additional days after the last dose of sotorasib and for at least 6 months afterwards after the last dose of FOLFIRINOX or gem/nab-P) or having a partner who is using a highly efficient method of contraception as described above
4. Pathologically confirmed treatment-naïve of advanced pancreatic adenocarcinoma harboring KRAS p.G12C mutation assessed by means of a IVDR compliant test).
5. Measurable disease per RECIST 1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Life expectancy > 3 months, in the opinion of the investigator.
8. Adequate hematologic, renal and hepatic organ function, defined as the following within 10 days prior study inclusion:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (without granulocyte colony-stimulating factor support within 2 weeks of laboratory test used to determine eligibility)
   * Hemoglobin ≥ 9.0 g/dL (without transfusion within 2 weeks of laboratory test used to determine eligibility)
   * Platelet count ≥ 100 x 109/L (without transfusion within 2 weeks of laboratory test used to determine eligibility)
   * Aspartate aminotransferase (AST) and ALT ≤ 2.5 times the upper limit of normal (ULN) or ≤5 times if liver metastasis
   * Serum bilirubin ≤ 1.5 x ULN
   * International normalized ratio (INR) ≤ 1.5 x ULN. Prothrombin time (PT) ≤ 1.5 x ULN may be used instead of INR for sites whose laboratory do not report INR
   * Creatinine clearance ≥ 30 mL/min (estimated by Cockcroft-Gault equation)
9. Ability to take oral medications and willing to record daily adherence to investigational product.

Exclusion Criteria:

1. Known history or positive viral test for human immunodeficiency virus (HIV).
2. Patients with known active hepatitis (i.e., Hepatitis B or C)

   * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible
   * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
3. Female: currently pregnant or breast-feeding or who plan to breastfeed while on study though 7 additional days after the last dose of sotorasib and for at least 6 months afterwards after the last dose of FOLFIRINOX or gem/nab-P
4. Myocardial infarction within 6 months of study Day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or cardiac arrhythmia requiring medication
5. Prior anti-tumor treatment for metastatic or advanced pancreatic adenocarcinoma*. Prior chemotherapy or radiotherapy in the adjuvant or neoadjuvant setting is acceptable if received > 6 months prior to study enrolment

   *If initiation of treatment is deemed urgent by the investigator, patients can receive 1st month of Standard of Care (SoC) gem/nab-P (1 cycle) or FOLFIRINOX (2 cycles) during screening. This first month of gem/nab-P or FOLFIRINOX is not a requirement of the study and is not part of this clinical study
6. Active infection requiring antibiotics within 1 weeks of study enrollment.
7. Other malignancy unless curatively treated with no evidence of disease for ≥2 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, and/or ductal carcinoma in situ.
8. Significant gastrointestinal disorder that results in significant malabsorption, requirement for IV alimentation, or inability to take oral medication.
9. History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis.
10. Presence of any condition that, in the opinion of the investigator, renders the patient at high risk from treatment complications or might affect the interpretation of the results of the study.
11. Significant uncontrolled concomitant disease that could affect compliance with protocol procedures or interpretation of results or that pose a risk to patient safety, in the opinion of the investigator.
12. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures at a frequency greater than monthly. Patients with PleurX catheters or intraperitoneal drainage catheters in place may be considered for the study with Medical Monitor approval.
13. Major surgery within 4 weeks of study Day 1
14. Prior/concomitant therapy:

    * Previous treatment with a KRASG12C inhibitor
    * Use of warfarin. Other anticoagulation may be allowed
    * Use of known cytochrome P450 (CYP) 3A4 sensitive substrates and P-glycoprotein (P-gp) substrates (with a narrow therapeutic window), within 14 days or 5 half-lives of the drug or its major active metabolite, whichever is longer, prior to study Day 1 (see examples of sensitive substrates and P-glycoprotein substrates in Appendix A)
    * Use of strong inducers of CYP3A4 within 14 days or 5 half-lives (whichever is longer) prior to study Day 1 (see examples of strong inducers of CYP3A4 in Appendix A)
15. Patient has known sensitivity to any of the products or components to be administered during the study.
16. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of sotorasib combined with first-line chemotherapy for advanced pancreatic adenocarcinoma harboring KRAS p.G12C mutation. | 60 months
  Incidence of treatment-emergent adverse events (TEAEs) and related TEAEs (TRAEs) according to CTCAE V5.0.

SECONDARY OUTCOMES:
To evaluate the progression-free survival assessed by CT or MRI using RECIST 1.1 criteria of first-line chemotherapy combined with sotorasib for advanced pancreatic adenocarcinoma harboring KRAS p.G12C mutation | 60 months
  Progression-Free Survival (PFS) is defined as time from the first day of the study treatment (Day 1) until disease progression or death from any cause, whichever occurs first, for all patients, according to the investigator criteria.
To evaluate the overall survival of first-line chemotherapy combined with sotorasib for advanced pancreatic adenocarcinoma harboring KRAS p.G12C mutation. | 60 months
  The overall survival (OS) is defined as time from Day 1 until death from any cause.
Overall response (OR) | 60 months
  The overall response (OR) is defined as the best overall response complete response (CR) or partial response (PR), assessed per RECIST 1.1.
Disease control (DC) | 60 months
  The disease control (DC) is defined as the best overall response of CR or PR or of stable disease.
Duration of response (DOR) | 60 months
  The duration of response (DOR) is defined as the time from onset of response to progression or death due to any reason, whichever occurs earlier.
Duration of stable disease | 60 months
  The duration of stable disease is defined as the time from first disease control to disease progression per RECIST 1.1 criteria or death (due to any cause). For patients with disease control who have not progressed or died at last observation, duration of disease control will be censored at their last evaluable disease assessment date.

CONTACTS AND LOCATIONS:
Locations (25):
- France (10):
  - Sainte Catherine - Institut Avignon Provence, Avignon, France
  - Chu Besançon - Hôpital Jean Minjoz, Besançon, France
  - Chu Brest - Hôpital Morvan, Brest, France
  - Chu de Lille - Claude Huriez, Lille, France
  - Hôpital Léon Berard, Lyon, France
  - Chu Bordeaux - Hôpital Haut Lévêque, Pessac, France
  - Chu Poitiers, Poitiers, France
  - Chu Reims - Hôpital Robert Debré, Reims, France
  - Chu Toulouse, Toulouse, France
  - Hôpital Paul-Brousse, Villejuif, France
- Spain (15):
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitari Vall D'Hebron, Barcelona, Barcelona
  - Institut Català D'Oncologia L'Hospitalet (Ico), Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Donostia-Donostia Unibertsitate Ospitalea, Donostia / San Sebastian, Guipúzcoa
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Complejo Hospitalario Regional de Málaga, Málaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Complexo Hospitalario Universitario de Ourense, Ourense, OURENSE
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Salamanca, Salamanca, SALAMANCA
  - Hospital General Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No